CLINICAL TRIAL: NCT05823259
Title: The Impact of a Widely Accessible Respiratory Muscle Training Program Integrated with Patient Education Utilizing a Hybrid Telehealth Platform on Patient-Reported Constipation Outcome Scores: a Call to Treat Beyond the Pelvic Floor
Brief Title: The Impact of Respiratory Muscle Training and Patient Education on Chronic Constipation Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Lawrence Cahalin, Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230123
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Constipation; Constipation - Functional; Dyssynergia
Keywords: Pelvic floor dysfunction; Dyssynergic defecation
MeSH Terms: conditions — Constipation; Ataxia | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid Telehealth Inspiratory and Expiratory Muscle Training Program with Patient Education (Experimental): Participants will be instructed in performing a home respiratory muscle training program using a device called the Breather that trains both inspiratory and expiratory muscle strength for 8 weeks. They will also be provided patient education on proper breathing techniques to pass a bowel movement and optimal toilet posture.
  Interventions: Other: Hybrid Telehealth Program: Respiratory Muscle Training and Patient Education
- Standard of Care Physical Therapy With No Study Intervention (Active Comparator): A historical control group of participants who received about 8 weeks of standard physical therapy care that includes interventions such as biofeedback treatment, manual therapy, therapeutic exercise, and education on improving bowel health.
  Interventions: Other: Standard Physical Therapy Care

INTERVENTIONS:
Other: Hybrid Telehealth Program: Respiratory Muscle Training and Patient Education — A testing session will be held where subjects will undergo respiratory muscle testing using the Pro2Fit device to measure PIMax and PEmax. During this session, subjects will be instructed in a respiratory muscle training home program utilizing a provided device call the Breather. They will be instructed to perform this program consisting of breathing exercises for 2 sets of 10 repetitions, twice a day at a difficulty level of 5-7 on the Visual Analogue Scale (VAS) scale for 8 weeks. Subjects will be shown how to follow a training program every day utilizing the free companion application to the device "Breather Coach." If subjects have issues with using technology, they will be provided a physical log to record when they complete sessions. Ten to fifteen-minute Zoom sessions with the study coordinator will be held once a week to check in on how the program is progressing, compliance, and if the resistance can be increased.
  Arms: Hybrid Telehealth Inspiratory and Expiratory Muscle Training Program with Patient Education
Other: Standard Physical Therapy Care — A group of patients who receive standard physical therapy care for chronic constipation at the University of Miami that consists of biofeedback therapy, manual therapy, therapeutic exercise, and patient education.
  Arms: Standard of Care Physical Therapy With No Study Intervention

SUMMARY:
The primary aim of this study will be to determine if a respiratory muscle training program that includes both inspiratory muscle training (IMT) and expiratory muscle training (EMT), targeted at improving respiratory muscle performance-based measures combined with patient education about breathing on the toilet will improve patient satisfaction scores in individuals with chronic constipation (CC).

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Complaint of CC and associated symptoms
* Willing and able to sign an informed consent
* The ability to comply with study guidelines
* Report two or more of the following: straining during more than 25% of defecations, lumpy or hard stools more than 25% of defecations, sensations of incomplete bowel evacuation more than 25% of defecations, manual maneuvers to facilitate more than 25% of defecations, sensation of anorectal obstruction/blockage more than 25% of defecations, and fewer than 3 small bowel movements per week.

Exclusion Criteria:

* Rectal prolapse greater than grade 2
* Pregnancy
* Cognitive impairments
* Currently receiving physical therapy treatment for conditions associated with pelvic floor muscle dysfunction
* Recent surgery within the past 3 months without clearance from a medical doctor
* Medication usage that would interfere with their ability to exercise safely
* Individuals recovering from a confirmed eating disorder
* Recent unexplained weight loss >10lbs within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Change In Patient Assessment of Constipation Symptoms (PAC-SYM) | Baseline, 4 weeks, and 8 weeks
  The PAC-SYM questionnaire is a 12 item questionnaire that consists of three subscales: abdominal, rectal, and stool. Each item is scored 0-4 (0: Absent, 1: Mild, 2: Moderate, 3: Severe, 4: Very Severe). The final score is the average of the summed score divided by the number of items, ranging from 0: Absent, 1: Mild, 2: Moderate, 3: Severe, 4: Very Severe. A total raw score can range for 0-48, however the average score is used to indicate the level of constipation from 0-4 with a higher number indicating higher severity of constipation.

SECONDARY OUTCOMES:
Change In Maximal Inspiratory Pressure (PImax) | Baseline and 8 weeks
  PImax will be measured via the test of incremental respiratory endurance (TIRE) using the Pro2fit device and application. Values will be presented in cmH20. Minimal score will be a 0 with a higher value indicating greater inspiratory muscle strength.
Change In Maximal Expiratory Pressure (PEmax) | Baseline and 8 weeks
  PEmax will be measured via the test of incremental respiratory endurance (TIRE) using the Pro2fit device and application. Minimal score will be a 0 with a higher value indicating greater expiratory muscle strength.
Change in Hospital Depression and Anxiety Scale (HADS) | Baseline and 8 weeks
  Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with two subscales, each consisting of 7 items. For both subscales, scores between 8-10 indicate mild depression or anxiety, and scores in the range of 11-21 are indicative of depression or anxiety disorder. A cutoff score for both the anxiety and depression subscale of the HADS of ≥ 8 has been suggested as optimal in identifying depression and anxiety in individuals with irritable bowel syndrome (IBS), a disorder of gut-brain interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Cahalin, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No